CLINICAL TRIAL: NCT06006520
Title: Investigation of the Effects of Aerobic and Oropharyngeal Exercises on Sleep Quality in Patients With Obstructive Sleep Apnea Syndrome.
Brief Title: Effects of Exercise on Sleep Quality in Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar60
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Osa Syndrome
Keywords: OSAS; quality of life; sleep
MeSH Terms: conditions — Carnevale syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: oropharyngeal exercises and aerobic exercises
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): No exercises will be given.
  Interventions: Other: control
- oropharyngeal (Experimental): oropharyngeal exercises will be given.
  Interventions: Other: oro-granary exercises.
- aerobic (Experimental): In addition to oropharyngeal exercises, 50 minutes of moderate-intensity aerobic exercise will be given at least 3 days a week.
  Interventions: Other: oro-granary exercises.; Other: aerobic exercises

INTERVENTIONS:
Other: control — No exercises will be given.
  Arms: control group
Other: oro-granary exercises. — soft palate exercises language exercises facial exercises stomatognathic functions swallowing and chewing exercises
  Arms: aerobic; oropharyngeal
Other: aerobic exercises — We can think of aerobic exercise as a low-intensity long-term activity using large muscle groups (between 60-80% of maximal heart rate). For example; It includes activities such as walking, cycling, jogging, aerobic dancing, swimming.
  Arms: aerobic

SUMMARY:
the investigators aim in this study is to investigate the effects of aerobic and oropharyngeal exercises on sleep quality in patients with Obstructive Sleep Apnea Syndrome (OSAS).

DETAILED DESCRIPTION:
The study will be conducted in a randomized controlled manner. Participants will be divided into groups of 3 equal numbers using the simple randomization method. The control group will not be given exercise. The first intervention group will be given 10-15 minutes of oropharyngeal exercises. In addition to oropharyngeal exercises, the second intervention group will be given 50 minutes of moderate-intensity aerobic exercise at least 3 days a week. Both intervention groups will apply the given exercise program for 8 weeks. All participants will be evaluated 3 times in total, at the beginning of the treatment, at the 4th week and at the 8th week. Epworth Sleepiness Scale, Pittsburgh Sleep Quality Questionnaire, Fatigue Severity Scale, Berlin Questionnaire, 6-minute walk test, Modified Medical Research Council (MMRC) Dyspnea Scale, Functional Results of Sleep Scale (FOSQ) tests will be applied to the participants. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* People who want to participate in the study voluntarily
* People who do not regularly engage in physical activity
* Persons diagnosed with OSAS in the neurology outpatient clinic
* People between the ages of 18-57
* Apnea Hypopnea Index 15-30

Exclusion Criteria:

* Chronic obstructive pulmonary disease, presence of lung disease that may cause respiratory failure
* -Severe cardiac disease, congestive heart failure, detection of ejection fraction in echocardiography, uncontrollable cardiac ischemia
* History of previous cerebrovascular disease
* Neuromuscular disease
* Presence of periodic leg movements
* Serious medical illness or planned surgical intervention
* Psychiatric illness, substance abuse

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | 10 weeks
  It is used to measure the general sleepiness of people during the day. In Epworth Sleepiness Scale, 4 ratings are made for a total of 8 questions. The total score was 24, and more than 10 points were considered as daytime sleepiness.
Pittsburgh Sleep Quality Survey | 10 weeks
  The scale includes a total of 24 questions. 19 of these questions are self-evaluation questions, and 5 of them are answered by the individual's spouse or a roommate. These 5 questions are used for clinical information only and are not included in the scoring. The scale questions that determine sleep quality include various factors related to sleep quality. These questions are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems; 18 items were grouped as 7 component scores. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. The scale does not indicate the presence of sleep disorders or the prevalence of sleep disorders. However, it is stated that a total score of 5 and above indicates poor sleep quality.
Fatigue Severity Scale | 10 weeks
  The person indicates how much he or she agrees with each item by choosing numbers from 1 to 7. 1 means completely disagree, 7 means completely agree. The score range of the scale, which consists of 9 questions in total, is 9-63. A score of 36 or higher indicates severe fatigue.
Berlin Survey | 10 weeks
  It is a questionnaire consisting of questions about snoring, daytime sleepiness, and high blood pressure, which have been shown to be risk factors for sleep apnea in previous sleep studies. Presence of snoring more than 3-4 times a week, presence of witnessed sleep apnea, daytime sleepiness more than 3-4 times a week and presence of at least two of the conditions were considered risky for sleep apnea syndrome.
Functional Outcomes of Sleep Scale (FOSQ) | 10 weeks
  It is a test used to evaluate the physical, social and mental effects of excessive daytime sleepiness on daily life activities. In the Turkish version of the FOSQ, questions about sexual activities are excluded and it consists of 26 questions. Each question is evaluated as no difficulty, mild, moderate, extreme and scored between 0-4 points. Calculation of low scores in total indicates functional disability. Turkish validity and reliability have been demonstrated.

CONTACTS AND LOCATIONS:
Overall Officials: Eda ARSLAN, Study Chair — Uskudar University
Locations (1):
- Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JJ, Sundar KM. Evaluation and Management of Adults with Obstructive Sleep Apnea Syndrome. Lung. 2021 Apr;199(2):87-101. doi: 10.1007/s00408-021-00426-w. Epub 2021 Mar 13. PMID 33713177
- [Background] Chwiesko-Minarowska S, Minarowski L, Kuryliszyn-Moskal A, Chwiesko J, Chyczewska E. Rehabilitation of patients with obstructive sleep apnea syndrome. Int J Rehabil Res. 2013 Dec;36(4):291-7. doi: 10.1097/MRR.0b013e3283643d5f. PMID 23873222
- [Background] Mohammadi H, Aarabi A, Rezaei M, Khazaie H, Brand S. Sleep Spindle Characteristics in Obstructive Sleep Apnea Syndrome (OSAS). Front Neurol. 2021 Feb 25;12:598632. doi: 10.3389/fneur.2021.598632. eCollection 2021. PMID 33716919
- [Background] Xanthopoulos MS, Berkowitz RI, Tapia IE. Effects of obesity therapies on sleep disorders. Metabolism. 2018 Jul;84:109-117. doi: 10.1016/j.metabol.2018.01.022. Epub 2018 Feb 1. PMID 29409812
- [Background] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106
- [Derived] Arslan E, Sevgin O. The effects of Aerobic and oropharyngeal exercises on sleep quality of patients with obstructive sleep Apnoea syndrome: a randomized controlled study. Sleep Breath. 2024 Dec;28(6):2729-2736. doi: 10.1007/s11325-024-03157-3. Epub 2024 Sep 20. PMID 39302514